CLINICAL TRIAL: NCT00094497
Title: First International Randomized Trial in Locally Advanced and Metastatic Adrenocortical Carcinoma Treatment
Brief Title: Trial in Locally Advanced and Metastatic Adrenocortical Carcinoma Treatment (FIRM-ACT)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Collaborative Group for Adrenocortical Carcinoma Treatment (Other)
Collaborators: German Federal Ministry of Education and Research (Other Government); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Martin Fassnacht, Co-PI, Collaborative Group for Adrenocortical Carcinoma Treatment
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CO-ACT-001; NCT00924144 (obsolete NCT alias)
Record Dates: First submitted 2004-10-19; First posted 2004-10-20 (Estimated); Results first posted 2016-09-21 (Estimated); Last update posted 2016-09-21 (Estimated); Status verified 2016-09

CONDITIONS: Carcinoma, Adrenal Cortical
MeSH Terms: conditions — Adrenocortical Carcinoma | interventions — Etoposide; Doxorubicin; Cisplatin; Streptozocin; Mitotane

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- EDP-M (Active Comparator): etopodide, doxorubicin, cisplatin and mitotane
  Interventions: Drug: Etoposide; Drug: Doxorubicin; Drug: Cisplatin; Drug: Mitotane
- Sz-M (Active Comparator): streptozotocin and mitotane
  Interventions: Drug: Streptozotocin; Drug: Mitotane

INTERVENTIONS:
Drug: Etoposide
  Arms: EDP-M
Drug: Doxorubicin
  Arms: EDP-M
Drug: Cisplatin
  Arms: EDP-M
Drug: Streptozotocin
  Arms: Sz-M
Drug: Mitotane

SUMMARY:
The purpose of this study is to determine whether treatment with etoposide, doxorubicin, cisplatin and mitotane (EDP/M) prolongs survival as compared to streptozotocin and mitotane (Sz/M) in patients with advanced adrenocortical carcinoma (ACC) whose disease is not amenable to complete surgical resection.

DETAILED DESCRIPTION:
The Firm-ACT trial is the first ever conducted randomized controlled phase III trial in adrenocortical carcinoma (ACC), a rare malignancy with poor prognosis. It will provide results leading to the establishment of an urgently needed gold standard chemotherapy regimen for patients with locally advanced or metastatic ACC. To this end the trial compares the two most promising drug combinations investigated in phase II trials, considered by the "International Consensus Conference on Adrenal Cancer" (Ann Arbor/USA, 2003) as valuable first line treatments for advanced ACC. The first regimen consists of etoposide, doxorubicin, cisplatin plus mitotane (EDP-M), the second regiment employs streptozotocin plus mitotane (Sz-M). Over a period of five years this international trial will include 300 patients with advanced ACC from different European countries. Blood mitotane concentrations will be monitored, aiming at drug levels between 14 - 20 mg/L. Patients not responding to the first line treatment will be switched to the alternative regimen. The primary objective of this trial is to investigate whether EDP-M given as first line treatment will prolong survival as compared to Sz-M. Secondary endpoints are quality of life, time to progression, best overall response rate and duration of response. In addition, the trial evaluates the role of reaching therapeutic mitotane serum concentrations for survival and tumour response and assesses the value of the two alternative treatment regimens as second line therapy in advanced ACC. Moreover, the FIRM-ACT trial will generate a lasting structural basis for successful future trials in ACC.

In a substudy of 40 patients a detailed analysis of the pharmacokinetics of oral mitotane will be analysed. Two different mitotane treatment regimens ("low dose" vs. "high dose") will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of adrenocortical carcinoma
* Locally advanced or metastatic disease not amenable to radical surgery resection (Stage III-IV)
* Radiologically monitorable disease
* ECOG performance status 0-2
* Life expectancy > 3 months
* Age ≥18 years
* Adequate bone marrow reserve (neutrophils > 1500/mm3 and platelets > 100,000/mm3)
* Effective contraception in pre-menopausal female and male patients
* Patient's written informed consent
* Ability to comply with the protocol procedures (including availability for follow-up visits)
* Previous palliative surgery, radiotherapy or radiofrequency ablation is acceptable as long as radiologically monitorable disease is verifiable afterwards.

Exclusion Criteria:

* History of prior malignancy, except for cured non-melanoma skin cancer, curatively in situ cervical carcinoma, or other cancers treated with no evidence of disease for at least five years.
* Previous cytotoxic chemotherapy for adrenocortical carcinoma
* Renal insufficiency (serum creatinine ≥2 mg/dl or creatinine clearance ≤ 50 ml/min)
* Hepatic insufficiency (serum bilirubin ≥2 x the institutional upper limit of normal range and/or serum transaminases ≥ 3 x the institutional upper limit of normal range; exception: in patients on mitotane, transaminase levels up to 5 x the institutional upper limit of normal range are acceptable)
* Pregnancy or breast feeding
* Known hypersensitivity to any drug included in the treatment protocol
* Presence of active infection
* Any other severe clinical condition that in the judgment of the local investigator would place the patient at undue risk or interfere with the study completion
* Decompensated heart failure (ejection fraction <50%), myocardial infarction or revascularization procedure during the last 6 months, unstable angina pectoris, and uncontrolled cardiac arrhythmia
* Current treatment with other experimental drugs and/or previous participation in clinical trials with other experimental agents for adrenocortical carcinoma
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 304 (Actual)
Dates: Start 2004-06; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Britt Skogseid, MD, Study Chair — Uppsala University Hospital; Martin Fassnacht, MD, Principal Investigator — University of Würzburg
Locations (32):
- United States (2):
  - National Cancer Institute - Center for Cancer Research, Bethesda, Maryland
  - University of Michigan, Department of Internal Medicine, Ann Arbor, Michigan
- Royal Adelaide Hospital, Adelaide, Australia
- University of Graz, Graz, Austria
- France (6):
  - Clinique Marc Linquette, Lille
  - Centre Leon Berard, Lyon
  - Hospital de Marseille la timone, Marseille
  - Cochin Hospital, Paris
  - Hospital Bordeaux haut leveque, Pessac
  - Institut Gustave Roussy, Villejuif
- Germany (10):
  - Charité-University, Dept. of Endocrinology; Campus Benjamin Franklin, Berlin
  - Charité-Universitätsmedizin Berlin - Campus Mitte, Berlin
  - Dept. of Medicine III, Dresden
  - University of Duesseldorf, Dept. of Endocrrinology, Düsseldorf
  - Zentrum für Innere Medizin - Endokrinologie des Universitätsklinikum Essen, Essen
  - Endokrinologie Medizinische Hochschule Hannover, Hanover
  - Otto-von-Guericke University; Dept. of Endocrinology, Magdeburg
  - Dept of Medicine I, Mainz
  - University of Munich, Dept. of Internal Medicine (Innenstadt), Munich
  - University of Wuerzburg - Dept. of Medicine, Würzburg
- Italy (2):
  - University of Turin, Dept of Internal Medicine, Orbassano
  - Clinica Endocrinologica, Università di Padova, Azienda Ospedaliera di Padova, Padua
- Netherlands (5):
  - Vrije Universiteit Medisch Centrum, Amsterdam
  - Academisch Medisch Centrum; Dept. of Endocrinology, Amsterdam
  - Maxima Medisch Centrum; Dept. of Internal Medicine, Eindhoven
  - University Hospital Groningen; Dept. of Internal Medine, Groningen
  - Leiden University Medical Center, Leiden
- Sweden (5):
  - Department of Oncology, Sahlgrenska University Hospital, Gothenburg
  - Department of Oncology, Linköping University Hospital, Linköping
  - Department of Medicine, The Jubileum Institute, Lund University, Lund
  - Dept of Surgery, Karolinska Hospital, Stockholm, Stockholm
  - Uppsala University Hospital - Dept of Medical Sciences, Uppsala

REFERENCES:
- [Result] Fassnacht M, Terzolo M, Allolio B, Baudin E, Haak H, Berruti A, Welin S, Schade-Brittinger C, Lacroix A, Jarzab B, Sorbye H, Torpy DJ, Stepan V, Schteingart DE, Arlt W, Kroiss M, Leboulleux S, Sperone P, Sundin A, Hermsen I, Hahner S, Willenberg HS, Tabarin A, Quinkler M, de la Fouchardiere C, Schlumberger M, Mantero F, Weismann D, Beuschlein F, Gelderblom H, Wilmink H, Sender M, Edgerly M, Kenn W, Fojo T, Muller HH, Skogseid B; FIRM-ACT Study Group. Combination chemotherapy in advanced adrenocortical carcinoma. N Engl J Med. 2012 Jun 7;366(23):2189-97. doi: 10.1056/NEJMoa1200966. Epub 2012 May 2. PMID 22551107
- See also: Click here for more information about this study: First International Randomized trial in locally advanced and Metastatic Adrenocortical Carcinoma Treatment (FIRM-ACT) — http://www.firm-act.org

RESULTS

PARTICIPANT FLOW:
Groups:
- EDP-M: etopodide, doxorubicin, cisplatin and mitotane
  Etoposide
  Doxorubicin
  Cisplatin
  Mitotane
  participants who progressed during first line therapy, were eligible to the alternative treatment (Sz-M)
- Sz-M: streptozotocin and mitotane
  Streptozotocin
  Mitotane
  participants who progressed during first line therapy, were eligible to the alternative treatment (EDP-M)
Period: Overall Study
Arm/Group | EDP-M | Sz-M
Started | 151 | 153
Treated | 148 | 149
Received Second Line Therapy | 84 | 101
Completed | 151 | 153
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | EDP-M | Sz-M | Total
Number analyzed (Participants) | 151 | 153 | 304
Age, Customized [Number; unit: participants]
  >= 18 years | 151 | 153 | 304
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 91 | 92 | 183
  Male | 60 | 61 | 121
tumor stage [Number; unit: participants]
  III | 0 | 1 | 1
  IV | 151 | 152 | 303
ECOG [Number; unit: participants] — Eastern Cooperative Oncology Group performance status score (ranges from 0, asymptomatic - 5, dead)
  participants
    0 | 73 | 72 | 145
    1 | 64 | 60 | 124
    2 | 13 | 21 | 34
    4 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: participants who died among those randomized to first-line therapy
Time Frame: every 8 weeks until death up to 5 years
Measure: Number; unit: participants
Arm/Group | EDP-M | Sz-M
Number analyzed (Participants) | 151 | 153
participants | 108 | 124

2. Secondary Outcome: Progression-free Survival
Time Frame: every 8 weeks until progression or death up to 5 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | EDP-M | Sz-M
Number analyzed (Participants) | 151 | 153
months | 5.0 [3.5 to 6.9] | 2.1 [2.04 to 2.33]

3. Secondary Outcome: Change in Quality of Life as Measured by QLQ-C30
Description: scale ranged from 0 to 100 with higher score meaning greater quality of life
Time Frame: baseline and 8 weeks
Population: participants with data on both time points
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | EDP-M | Sz-M
Number analyzed (Participants) | 60 | 39
units on a scale | -6.0 (21.4) | -7.7 (25.6)

4. Secondary Outcome: Best Overall Response Rate
Description: RECIST 1.0 was used to evaluate response
Time Frame: every 8 weeks up to 5 years
Measure: Number; unit: participants
Arm/Group | EDP-M | Sz-M
Number analyzed (Participants) | 151 | 153
participants
  complete response | 2 | 1
  disease-free by time of surgery | 4 | 2
  partial response | 29 | 11
  stable disease | 53 | 34
  progressive disease | 43 | 88
  did not receive treatment | 3 | 4
  could not be evaluated | 17 | 13

5. Secondary Outcome: Number of Disease-free Patients
Description: complete response or disease-free by time of surgery
Time Frame: every 8 weeks until progression (up to 5 years)
Measure: Number; unit: participants
Arm/Group | EDP-M | Sz-M
Number analyzed (Participants) | 151 | 153
participants | 6 | 3

6. Other Pre Specified Outcome: TTP of Both Regimens as Second Line Treatment in Case of Failure of the Other Initial Regime
Time Frame: every 8 weeks until progression or until Dec 2010
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Pharmakinetics of Mitotane (Substudy)
Description: To study the relationship between mitotane dose (daily and cumulative) and mitotane plasma concentrations using one of two pre-defined treatment regimens (high-dose and low-dose).
Time Frame: 11 time points in the first 12 weeks
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Impact of Reaching Mitotane Blood Levels Between 14-20 mg/l in Both Arms on Survival and Overall Response Rate
Time Frame: every 8 weeks until progression or until Dec 2010
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: up to 5 years
Description: Other non-serious adverse events were not reliably collected and therefore not reported
Arm/Group | EDP-M | Sz-M
Serious Adverse Events (participants affected / at risk) | 86/148 | 62/149
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | EDP-M (N=148) | Sz-M (N=149)
adrenal insufficiency (Endocrine disorders) | 5 | 1
bone marrow toxicity (Blood and lymphatic system disorders) | 17 | 3
cardiovascular or thromboembolic events (Vascular disorders) | 10 | 0
fatigue or general health deterioration (General disorders) | 8 | 7
gastrointestinal disorder (Gastrointestinal disorders) | 6 | 12
impaired liver function (Hepatobiliary disorders) | 0 | 7
impaired renal function (Renal and urinary disorders) | 1 | 6
infection (Infections and infestations) | 10 | 4
neurologic toxicity (Nervous system disorders) | 5 | 4
respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 9 | 5
Other (General disorders) | 15 | 13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No